CLINICAL TRIAL: NCT02054793
Title: Phase Ib/II Study Evaluating Orteronel (Without Prednisone) Combined With Itraconazole In Men With Castration-Resistant Prostate Cancer (CRPC)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was never able to open due to lack of funding from the pharmaceutical company.
Sponsor: Emmanuel Antonarakis, MD (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Emmanuel Antonarakis, MD, Sponsor-Investigator, Johns Hopkins University
Organization: Johns Hopkins University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Itraconazole/Orteronel
Record Dates: First submitted 2014-01-30; First posted 2014-02-04 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Prostate Cancer; Castration-resistant Prostate Cancer
Keywords: metastatic disease; non-metastatic disease; prostate cancer; castration-resistant prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Itraconazole; orteronel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Itraconazole — 100 mg 200 mg 300 mg
  Other Names: Sporanox
Drug: Orteronel — 300 mg
  Other Names: TAK 700

SUMMARY:
This research is being done to test the safety and anti-cancer activity of the combination of an investigational drug called orteronel, with a drug called itraconazole in the treatment of castration-resistant prostate cancer.

Orteronel is an investigational drug known as a 17,20-lyase enzyme inhibitor, meaning that it blocks the formation of male sex hormones.

Itraconazole is approved by the Food and Drug Administration (FDA) for the treatment of various fungal infections such as fingernail/toenail infections and other more serious fungal infections. While it has shown evidence of activity against prostate cancer in prior studies, it is not approved for use in cancer. The FDA is allowing the use of orteronel and itraconazole in this research study. In addition to its antifungal properties, itraconazole was discovered to function to block angiogenesis (blood vessel formation to tumors) to block a cellular pathway thought to be important in prostate cancer known as the Hedgehog pathway.

Investigators hypothesize that blocking male sex hormone production with orteronel will increase reliance on the Hedgehog pathway in prostate cancer cells which can then be blocked with itraconazole and that the combination of these two drugs will be more effective than either alone.

DETAILED DESCRIPTION:
Hedgehog (Hh) pathway signaling may be important in prostate cancer progression and this pathway is upregulated in the castration-resistant state. More potent (maximal) castration achievable by CYP17 inhibition, using orteronel, may further upregulate Hh pathway activation. Itraconazole administered at high doses (600 mg/day) may function as a modest Hh inhibitor. In a pilot phase II trial, investigators have shown that single-agent high-dose itraconazole produced PSA reductions in 29% of men with metastatic castration-resistant prostate cancer (CRPC), reduced circulating tumor cell counts in 62% of patients with unfavorable baseline counts, and prolonged progression-free survival compared to historical data. Moreover, clinical responses to itraconazole appeared to correlate with Hh pathway suppression, as measured by GLI1 mRNA analysis from serial skin biopsies.

Investigators propose to evaluate the potent CYP17/lyase inhibitor, orteronel, in combination with itraconazole at escalating dose levels (100 mg BID, 200 mg BID, 300 mg BID) in men with non-metastatic or metastatic CRPC by conducting an open-label phase Ib/II trial. Importantly, unlike the related compound, ketoconazole, itraconazole very rarely results in adrenal suppression. Side effects previously seen at the highest dose of itraconazole (600 mg/day) were mild and included nausea, rash, diarrhea, vomiting, hypokalemia, edema, headache, hypertension, fever, pruritis, and abnormal liver function tests. Of note, orteronel will be given without concurrent prednisone in this trial. This is because the combination of itraconazole and corticosteroids can lead to Cushing's syndrome (hypercortisolism) by impairing corticosteroid metabolism through CYP3A4.

Therefore, this study provides an opportunity to evaluate a steroid-free orteronel combination regimen. If this combination is safe and tolerable, subsequent studies would aim to compare the clinical efficacy of orteronel-itraconazole versus orteronel alone using a randomized phase II trial design.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* must provide written consent
* must agree to use contraception
* has a diagnosis of castrate resistant prostate cancer
* normal clinical lab values ALT and AST must be ≤ 2.5 x the upper limit of normal (ULN). Total bilirubin must be ≤ 1.5 x ULN. Estimated creatinine clearance using the Cockcroft-Gault formula must be > 40 mL/minute Absolute neutrophil count (ANC) must be ≥ 1500/uL Platelet count must be ≥ 100,000/uL
* has stable medical conditions (including absence of acute exacerbations of chronic illnesses, serious infections or major surgery within 4 weeks before first dose of drug
* castrate level of testosterone (< 50ng/dL)
* screening calculated ejection fraction of > 50% by ECHO.

Exclusion Criteria:

* received prior therapy with orteronel, ketoconazole, aminoglutethimide, or abiraterone. Prior enzalutamide treatment is permitted.
* prior use of docetaxel for CRPC
* symptomatic metastatic disease with signs of rapid progression per investigator's clinical judgment or hepatic metastases
* currently receiving corticosteroids
* concurrent use of acid-lowering drugs (histamine antagonists, proton pump inhibitors)
* known hypersensitivity to compounds related to orteronel, orteronel excipients, itraconazole or related compounds including other azole antifungals
* concurrent administration of other drugs that significantly interact with CYP450 3A4 isoenzyme
* known brain metastases
* treatment with any investigational products within one month before the first dose of study drug
* diagnosis of or treatment for another systemic malignancy within 2 years before the first dose of study drug, or previously diagnosed with another malignancy and have any evidence of residual disease
* history of myocardial infarction, unstable symptomatic ischemic heart disease, ongoing arrhythmias of Grade >2 (NCI CTCAE version 4.0, effective dates 14 June 2010), thromboembolic events (e.g. deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events), or any other cardiac condition (e.g. pericardial effusion, restrictive
* has New York Heart Association (NYHA) Class III or IV heart failure
* uncontrolled hypertension despite appropriate medical therapy (systolic blood pressure >160 mm Hg or diastolic blood pressure >90 mmHg) at 2 separate measurements no more than 60 minutes apart during the Screening visit).
* has known gastrointestinal (GI) disease or GI procedure that could interfere with the GI absorption or tolerance of orteronel, including difficulty swallowing tablets
* likely unable to comply with the protocol or cooperate fully with the investigator and site personnel

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 12 months after study initiation
  This is a dose escalation phase I trial where 3 subjects will be enrolled at each dose level. If no dose limiting toxicities (DLTs) are seen at a dose level, the study moves to the next dose level. If 1 DLT is seen, 3 additional subjects must be enrolled at the current dose level. If 2-3 DLTs are seen, we will stop accrual to that particular dose level, and the previous dose level becomes the maximum tolerated dose.

SECONDARY OUTCOMES:
Grade and severity of adverse events | up to 25 months
  To determine the safety and tolerability of the combination regimen: orteronel + itraconazole. The grade and severity of adverse events will be assessed using CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: EMMANUEL ANTONARAKIS, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Johns Hopkins University, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan